CLINICAL TRIAL: NCT02126163
Title: Promoting Responsible Drinking: An Internet-based, Interactive Computer Tailored Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pro-Change Behavior Systems (Other)
Responsible Party: Principal Investigator, Deborah Levesque, Chief Science Officer, Pro-Change Behavior Systems
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2R44AA01733-02
Record Dates: First submitted 2014-04-27; First posted 2014-04-29 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Regular Heavy AOD Use; Excessive Drinking
Keywords: Excessive Drinking; Hazardous Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): The treatment group will receive three interactive Computer Tailored Intervention (CTI) sessions during the course of six months, which will include tailored feedback based on the user's responses, and two assessment only follow-up sessions at twelve and eighteen months.
  Interventions: Behavioral: Treatment Group
- Control Group (No Intervention): The control group will receive four assessment only sessions during 18 months.

INTERVENTIONS:
Behavioral: Treatment Group — Responsible Drinking intervention sessions include an internet-based, computer-tailored intervention (CTI) grounded in the Transtheoretical Model of Behavior Change (TTM). The intervention includes stage-matched and tailored feedback on alcohol use, alcohol-related problems, and theoretically identified behavior change strategies, as well as access to a web-based portal with stage-matched interactive activities to reinforce and promote stage progression. Finally, the intervention will include 7 months of stage-matched behavior change SMS messages.
  Arms: Treatment Group

SUMMARY:
Excessive alcohol use is associated with a range of serious and costly health, social, and economic consequences at the individual and societal level. This program of research serves as a venue by which to produce and test an innovative, science-based, and cost-effective means to intervene in a private, convenient, and individualized way with employed adults who report non-dependent levels of risky drinking. Responsible Drinking offers computer-tailored intervention sessions directed at increasing readiness to limit drinking to national guidelines for low-risk drinking and a complementary dynamic web portal providing additional information, activities, and strategies designed to activate and reinforce the change process. The primary objective is to complete and enhance the development of Responsible Drinking and test it in an effectiveness trial. In Phase II the program capabilities and innovation will expand to integrate the e-Health components (CTI and e-Workbook) with m-Health (mobile health) technologies. The e-Health components will be enhanced to offer a more interactive and engaging user experience. In addition, m-Health technologies (text messaging and mobile device browsing optimization) will be integrated to support engagement in the program and flexible delivery options. 996 employed adults will be recruited to participate in the randomized trial. The treatment group will receive three intervention sessions during the course of six months and group differences on a number of outcomes will be evaluated at 12 and 18 month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. 21 years of age or older
3. not enrolled full-time in college
4. employed part or full time
5. not pregnant
6. consumed alcohol in the past 30 days
7. exceeded the NIAAA gender-specific low-risk drinking guidelines in the last 30 days
8. not currently interested in or ever having received treatment for substance abuse or dependence
9. not ever having received a physician recommendation to avoid or reduce alcohol use
10. scoring 9 or less on the Alcohol Use Disorders Identification Test (AUDIT-C).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who reach criteria for limiting drinking according to low-risk drinking guidelines | 18 month follow-up
  To assess efficacy by comparing treatment and control group participants who are at-risk at baseline - assessed using a self-report Transtheoretical Model of Behavior Change (TTM) stage of change measure
Quantity of alcohol use (number of drinks per week, number of drinks per drinking day) | 18 month follow-up
  To assess efficacy by comparing treatment and control group participants who are at-risk at baseline - accessed using continuous measures of drinking behavior
Frequency of alcohol use (days drinking above recommended limits during the past month, number of drinking days in the past month) | 18 month follow-up
  To assess efficacy by comparing treatment and control group participants who are at-risk at baseline- accessed using continuous measures of drinking behavior

SECONDARY OUTCOMES:
Ratings of alcohol-related problems | 18 month follow-up
  To assess the efficacy of the intervention by comparing treatment and control group participants who are at-risk at baseline - accessed using the SIP measure
Well-being related to productivity | 18 month follow-up
  To assess the efficacy of the intervention by comparing treatment and control group participants who are at-risk at baseline - Accessed using WBA-F and WBA-P

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Levesque, Ph.D., Principal Investigator — Pro-Change Behavior Systems, Inc.
Locations (1):
- Pro-Change Behavior Systems, Inc., South Kingstown, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mauriello LM, Gokbayrak NS, Van Marter DF, Paiva AL, Prochaska JM. An Internet-Based Computer-Tailored Intervention to Promote Responsible Drinking: Findings from a Pilot Test with Employed Adults. Alcohol Treat Q. 2011 Winter;30(1):91-108. doi: 10.1080/07347324.2012.635528. PMID 22448087